CLINICAL TRIAL: NCT06118918
Title: Impact of Rehabilitation on Anxiety, Depression, Perceived Health Status, and Readmission Among Patients After Coronary Artery Bypass in Jordan
Brief Title: Effect of Cardiac Rehabilitation on Health Status, Emotional Outcomes, and 90-day Readmission Rate Among Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, ALI SULEIMAN HARBI, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9771044993
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Health Status; Anxiety; Depression; 90-day Readmission
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The interventional arm (participants who will received the cardiac rehabilitation program (Experimental): this arm will receive the cardiac rehabilitation program after completing the cardiac surgery and being assessed for eligibility.
  Interventions: Behavioral: Phase II comprehensive cardiac rehabilitation program
- the control arm (who will receive the usual care) (No Intervention): the control group will receive the usual care ( the usual instruction and general advice from the physicians and the nurses)

INTERVENTIONS:
Behavioral: Phase II comprehensive cardiac rehabilitation program — the program extends over 3 months after cardiac surgery. The program includes exercise, health education, and stress management. all content will be delivered to the participants through the WhatsApp application as instruction videos and short lectures. exercise will be gradually increased in terms of intensity, and duration. health education will cover topics like a healthy diet blood pressure, blood cholesterol control, smoking cessation …etc. stress management will include relaxation therapy, breathing control, behavioral change, and other strategies to control stress. Phone call follow-ups once weekly will be made by one of the research team to evaluate the adherence and answer potential questions All interventions are guided by universal guidelines like the Australian Cardiovascular Health and Rehabilitation Association (ACRA) and American Heart Association (AHA
  Arms: The interventional arm (participants who will received the cardiac rehabilitation program

SUMMARY:
this study aims to investigate the effect of the cardiac rehabilitation program on perceived health, status, anxiety, depression, and 90-day readmission rates for post-cardiac surgery patients. The participants in this study will be randomly allocated to either an experimental or control group, the experimental group will receive the cardiac rehabilitation programThe cardiac rehabilitation program extends over 3 months after cardiac surgery. The program includes exercise, health education, and stress management. All content will delivered to the participants through the WhatsApp application as instruction videos and short lectures. exercise will be gradually increased in terms of intensity, and duration. Health education will cover topics like a healthy diet blood pressure, blood cholesterol control, smoking cessation..etc. Stress management will include relaxation therapy, breathing control, behavioral change, and other strategies to control stress. All interventions are guided by universal guidelines like the Australian Cardiovascular Health and Rehabilitation Association (ACRA) and American Heart Association (AHA)..All potential participants will be assessed before being involved in the study. assessment including a general physical examination, inspection of the surgical site, and recent history for potential patient symptoms after discharge, such as chest pain, palpitation, fatigue, or dyspnea. The assessment includes electrocardiograph (ECG), blood samples, and echocardiography analyses. Based on the findings of this assessment, patients will be classified by the cardiologist as either grade I, II, III, or IV, according to the New York Heart Association (NYHA) Classification. Patients who will be eligible to participate in the present study should be grade I or II in the NYHA Classification for dyspnea. Participants in the control group will receive the usual care (general instructions and advice from physicians and nurses). All materials will be delivered to all participants after completing the study.

ELIGIBILITY:
Inclusion Criteria:

1. . aged over 18 years.
2. underwent cardiac surgery.
3. classified as grade I or II according to NYHA classification of dyspnea by the physician.
4. does not complain of any physical or mental condition preventing him or her from participating.
5. agree to participate in the study.

Exclusion Criteria:

1. aged under 18 years.
2. classified as grade III or IV according to NYHA classification of dyspnea by the physician.
3. complain of any physical or mental condition preventing him or her from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Perceived health status | At base-line, after 12 weeks , and 1 month later
  Short form-36 health survey will be used to measure the perceived health status..
  The score ranges from 0 to 100. A high score defines a more favorable health state.
Anxiety level | At base-line, after 12 weeks, and 1 month later
  Anxiety will be measured using the Hospital Anxiety and depression scale(HADS). The score ranges from 0 to 21. The highest score indicates worse symptoms.
Depression | At base-line, after 12 weeks , and 1 month later
  Depression will be measured using the Hospital anxiety and depression scale(HADS).
  The score ranged from 0 to 21. The highest score indicates worse symptoms.
90-day readmission rate | after90 days
  readmission rate will measured by reviewing patient medical record

CONTACTS AND LOCATIONS:
Overall Officials: ALI SU HARBI, Principal Investigator — University Putra Malaysia
Locations (1):
- Prince Hamzah hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD